CLINICAL TRIAL: NCT01176162
Title: PREMALDO : Aldosterone Resistance in Preterm Infants : Assessment by a Non Invasive Measurement of Urinary Aldosterone
Brief Title: Aldosterone Resistance in Preterm Infants
Acronym: PREMALDO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: P081211; B91017-20 (Other Grant/Funding Number: Proper Authorithies : AFSSaPS)
Record Dates: First submitted 2010-07-06; First posted 2010-08-05 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Newborn
Keywords: Non Invasive measurement; Preterm infants; Aldosterone resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Urinary samples will be collected onto a gauze compress, during the first 24 hours of life, at day three, and at 1, 3, 6 and 12 months.
  * A blood sample will be obtained from systematic umbilical cord blood collection at birth and during the Guthrie test at day three
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group "< 28": • Gestational Age < 28 weeks
- Group "28 - < 33": • Gestational Age : 28 - < 33 weeks
- Group "33- < 37": Gestational Age : 33- < 37 weeks
- Group "> 37": Gestational Age > 37 weeks

SUMMARY:
In the neonatal period, the human kidney is characterized by a functional immaturity responsible for an impaired ability to regulate water and sodium homeostasis, which is exacerbated by prematurity. This altered sodium handling could be related to a partial renal aldosterone resistance. Renal sodium reabsorption and potassium excretion are mainly controlled by aldosterone, after binding to the mineralocorticoid receptor (MR). The investigators have analyzed MR expression throughout human and mouse renal development, and the investigators found a weak MR expression at birth. The investigators have conducted a pilot study in full-term newborns, which confirmed a partial neonatal aldosterone resistance. This study also highlighted that urinary aldosterone is the best index to accurately assess aldosterone sensitivity at birth.

DETAILED DESCRIPTION:
Principal objective:

To assess aldosterone resistance at birth by a non invasive measurement of urinary aldosterone, in order to evaluate its intensity as a function of gestational age. Determination of normal values of urinary aldosterone concentration in each group.

Secondary objectives:

Comparison of plasma and urinary electrolytes concentrations with hormonal measurements and clinical parameters. Evolution of these biological parameters throughout the first year of life, depending on gestational age at birth.

Methodology : multicentric study, open study Two hundred-forty newborns will be included in order to constitute 4 groups of 60 children, classified according to their gestational age: < 28 GW, 28 - < 33 GW, 33- < 37 GW, > 37 GW.

Inclusion criteria: every newborn will be included, after written parental consent was obtained.

Study :

Urinary samples will be collected onto a gauze compress, during the first 24 hours of life, at day three, and at 1, 3, 6 and 12 months. A blood sample will be obtained from systematic umbilical cord blood collection at birth and during the Guthrie test at day three. Aldosterone and renin concentrations will be measured in BICETRE Hospital laboratory. Plasma and urinary electrolyte concentrations will be measured in the Biochemistry department. DNA samples will also be gathered from umbilical cord blood for future genetic investigations (functional polymorphisms of the MR gene).

Perspectives This study will permit to assess the intensity of aldosterone resistance in full-term and preterm newborns, by a non invasive method. It should bring new insights into the mechanisms of hormonal regulation of sodium balance in preterm newborns and during the first year of life. Urinary aldosterone assessments may open new perspectives for therapeutic management of water and sodium waste in premature infants.

ELIGIBILITY:
Inclusion criteria :

* Maternal

  * Maternal age ≥ 18 and ≤ 45 years,
  * Written parental consent
  * Normal obstetrical ultrasounds
* Neonatal - Birth by vaginal delivery or cesarean section

Exclusion criteria :

* Maternal

  * Type 1 or type 2 diabetes,
  * Adrenal or hypophyseal deficiency
  * Treatment for arterial hypertension
* Neonatal

  * Perinatal anoxia (defined by an Apgar score < 5 at 5 min and pH < 7,10 and lactacidemia > 9 mmol/l at blood cord).
  * Congenital malformation
  * Chromosomic abnormalities

Ages: 24 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Every newborn without congenital malformation will be included, after written parental consent was obtained
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
urinary aldosterone | during the first year of life
  Determination of normal values of urinary aldosterone concentration in each group (24 first hours, day three, and at 1 and 3 months)

SECONDARY OUTCOMES:
plasma electrolytes concentrations | first year of life
  Comparison of plasma and urinary electrolytes concentrations with hormonal measurements and clinical parameters. Evolution of these biological parameters throughout the first year of life, depending on gestational age at birth.
urinary electrolytes concentrations | first year of life
  Comparison of plasma and urinary electrolytes concentrations with hormonal measurements and clinical parameters. Evolution of these biological parameters throughout the first year of life, depending on gestational age at birth.
hormonal measurements | first year of life
  Comparison of plasma and urinary electrolytes concentrations with hormonal measurements and clinical parameters. Evolution of these biological parameters throughout the first year of life, depending on gestational age at birth.
clinical parameters | first year of life
  Comparison of plasma and urinary electrolytes concentrations with hormonal measurements and clinical parameters. Evolution of these biological parameters throughout the first year of life, depending on gestational age at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal BOILEAU, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Assistance Publique- Hôpitaux de Paris: Antoine Beclere Hospital, Clamart, Île-de-France Region, France

REFERENCES:
- [Background] Martinerie L, Viengchareun S, Delezoide AL, Jaubert F, Sinico M, Prevot S, Boileau P, Meduri G, Lombes M. Low renal mineralocorticoid receptor expression at birth contributes to partial aldosterone resistance in neonates. Endocrinology. 2009 Sep;150(9):4414-24. doi: 10.1210/en.2008-1498. Epub 2009 May 28. PMID 19477942
- [Derived] Martinerie L, Pussard E, Yousef N, Cosson C, Lema I, Husseini K, Mur S, Lombes M, Boileau P. Aldosterone-Signaling Defect Exacerbates Sodium Wasting in Very Preterm Neonates: The Premaldo Study. J Clin Endocrinol Metab. 2015 Nov;100(11):4074-81. doi: 10.1210/jc.2015-2272. Epub 2015 Sep 8. PMID 26348350